CLINICAL TRIAL: NCT00004274
Title: Controlled Study of Estrogen Effects on Cognitive and Social Function in Girls With Turner's Syndrome
Brief Title: Effect of Estrogen on Mental and Social Functioning in Girls With Turner's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Jefferson Medical College of Thomas Jefferson University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11680; TJU-11680
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Turner's Syndrome
Keywords: Turner's syndrome; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Turner Syndrome; Genetic Diseases, Inborn; Rare Diseases | interventions — Estrogens

INTERVENTIONS:
Drug: Estrogen

SUMMARY:
RATIONALE: Turner's syndrome is a disease in which females are missing all or part of one X chromosome and do not produce estrogen. Giving estrogen is standard treatment for girls who have Turner's syndrome. Estrogen may be effective treatment for mental and social functioning problems experienced by girls with Turner's syndrome.

PURPOSE: Clinical trial to study the effectiveness of long term estrogen therapy on mental and social functioning in girls who have Turner's syndrome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Participants are evaluated for cognitive and social function at entry and 4 years following entry. Assessments include the Wechsler Intelligence Scale for Children-Revised, a child behavior checklist, the Children's Self-Concept Scale, and visual-spatial, visual-motor, attention, memory, language, and facial recognition tasks.

Patients (and parents) undergo X-chromosome analysis; brain magnetic imaging is optional.

Controls are matched using school selection and telephone interviews.

A study duration of 12 years is estimated.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Girls aged 8 and 12 years with Turner's syndrome-compatible karyotype
* Age-matched girls without Turner's syndrome entered as controls
* Concurrent registration on Thomas Jefferson University growth study required of subjects with Turner's syndrome

Ages: 8 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260
Dates: Start 1990-02

CONTACTS AND LOCATIONS:
Overall Officials: Judith Levine Ross, Study Chair — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Jefferson Medical College of Thomas Jefferson University, Philadelphia, Pennsylvania, United States